CLINICAL TRIAL: NCT00544076
Title: Erectile Dysfunction Recovery in Men Age </=65 Treated With Bilateral Nerve Sparing Robotic Assisted Prostatectomy (BNS-RAP) for Prostate Cancer
Brief Title: ED Recovery in Men Age </=65 Treated With Bilateral Nerve Sparing Robotic Assisted Prostatectomy for Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Accrual too slow
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 04071; NCI-2009-01602 (Registry Identifier: NCI CTRP); CDR0000570272 (Registry Identifier: PDQ)
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Results first posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Prostate Cancer; Male Erectile Disorder; Stage I Prostate Cancer; Stage II Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — Sildenafil Citrate; Alprostadil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sildenafil Citrate/Mo+Aprostadil/day (Experimental): Patients receive intraurethral alprostadil once daily for up to 9 months in the absence of disease progression or unacceptable toxicity. Patients also receive 3 doses of oral sildenafil citrate at least 48 hours apart monthly for up to 18 months. Patients on all three arms will have undergone robotic-assisted laparoscopic surgery. All patients will take part in the questionnaire administration and quality-of-life assessments.
  Interventions: Drug: sildenafil citrate; Drug: alprostadil; Procedure: robotic-assisted laparoscopic surgery; Procedure: quality-of-life assessment; Other: questionnaire administration
- Sildenafil Citrate Monthly (Active Comparator): Patients receive 3 doses of oral sildenafil citrate on 3 separate occasions at least 48 hours apart monthly for 18 months. Patients on all three arms will have undergone robotic-assisted laparoscopic surgery. All patients will take part in the questionnaire administration and quality-of-life assessments.
  Interventions: Drug: sildenafil citrate; Procedure: robotic-assisted laparoscopic surgery; Procedure: quality-of-life assessment; Other: questionnaire administration
- Daily Sildenafil Citrate (Experimental): Patients receive oral sildenafil citrate once daily for up to 9 months in the absence of disease progression or unacceptable toxicity. Patients also receive 3 doses of oral sildenafil citrate at least 48 hours apart monthly for up to 18 months. Patients on all three arms will have undergone robotic-assisted laparoscopic surgery. All patients will take part in the questionnaire administration and quality-of-life assessments.
  Interventions: Drug: sildenafil citrate; Procedure: robotic-assisted laparoscopic surgery; Procedure: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Drug: sildenafil citrate — Given orally
  Other Names: Viagra
Drug: alprostadil — Given intraurethrally
  Other Names: Caverject; MUSE; PGE1; prostaglandin E1
  Arms: Sildenafil Citrate/Mo+Aprostadil/day
Procedure: robotic-assisted laparoscopic surgery — Undergo prostatectomy
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
RATIONALE: Sildenafil citrate and alprostadil may help patients who have undergone prostatectomy for prostate cancer to recover from erectile dysfunction.

PURPOSE: This randomized clinical trial is studying giving sildenafil together with alprostadil in treating patients undergoing nerve-sparing robotic-assisted radical prostatectomy for nonmetastatic prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of erectile function (defined as the ability to achieve and maintain an erection sufficient for intercourse without the use of pharmacological assistance) at 1 year post-operatively in men undergoing BNS-RAP without the use of post-operative maintenance pharmacotherapy.

II. To describe whether early post-operative maintenance pharmacotherapy Viagra can improve return of erectile function at 1 year post-operatively in patients undergoing BNS-RAP.

III. To describe if early post-operative maintenance pharmacotherapy Viagra can decrease the time-to-return of erectile function in patients undergoing BNS-RAP.

SECONDARY OBJECTIVES:

I. To describe whether early post-operative maintenance pharmacotherapy MUSE can improve return of erectile function at 1 year post-operatively in patients undergoing BNS-RAP.

II. To describe if early post-operative maintenance pharmacotherapy MUSE can decrease the time-to-return of erectile function in patients undergoing BNS-RAP.

III. To compare sexual function quality of life in men undergoing early post-operative maintenance pharmacotherapy to those without early post-operative maintenance pharmacotherapy.

IV. To compare the rate of potency at 1, 3, 6, 9, 12, and 18 months in men using Viagra versus MUSE for early post-operative maintenance pharmacotherapy.

V. To describe the dropout rate for MUSE maintenance pharmacotherapy secondary to urethral pain in men using 2% Lidocaine lubricant.

VI. To describe if penile length is decreased following BNS-RAP. VII. To describe if penile length at one year is different in men who have return of potency versus those with no return of potency.

OUTLINE: Patients receive 2 doses of intraurethral alprostadil prior to undergoing bilateral nerve-sparing robotic-assisted prostatectomy. Within 4 weeks after surgery, patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive intraurethral alprostadil once daily for up to 9 months in the absence of disease progression or unacceptable toxicity. Patients also receive 3 doses of oral sildenafil citrate at least 48 hours apart monthly for up to 18 months.

ARM II: Patients receive 3 doses of oral sildenafil citrate on 3 separate occasions at least 48 hours apart monthly for 18 months.

ARM III: Patients receive oral sildenafil citrate once daily for up to 9 months in the absence of disease progression or unacceptable toxicity. Patients also receive 3 doses of oral sildenafil citrate at least 48 hours apart monthly for up to 18 months.

After completion of study treatment, patients are followed periodically for up to 18 months.

ELIGIBILITY:
Inclusion Criteria

* All patients undergoing BNS-RAP for prostate cancer will be asked to participate
* Ability to achieve erections sufficient for intercourse prior to surgery and an SHIMS-5 score of >= 22
* Must maintain follow up care at COH for visits 1, 3, 6, 9, 12, and 18 months post surgery
* Participants willing to participate on study for a minimum of 18 months
* Consented participant on the Prostate database study (protocol 00149)
* Patients must have a clinical stage of < T3
* Gleason score < 8 on post-operative pathological sample prior to randomization

Exclusion Criteria

* Metastatic disease
* Coronary artery disease on nitrate therapy (including oral sublingual nitrates)
* Unable to maintain follow up visits at COH at 1, 3, 6, 9, 12, and 18 months post-operatively
* Pathology diagnosis >= pT3
* Prior hormonal treatment use for prostate cancer or low serum testosterone
* Allergy to prostaglandin PGE1, Lidocaine, or Viagra
* Gleason score >= 8 on post-operative pathological sample prior to randomization
* Concomitant use of cytochrome P450 3AY inhibitors (cimetidine, erythromycin, ketoconazole, or protease inhibitors)
* SHIMS-5 score =< 21

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Crocitto, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 patients were not randomized, for the following reasons:
  1. ineligible upon surgery - 4 patients
  2. patient withdrew or not returning to COH - 2 patients
  3. did not have BNS procedure -- 2 patients
  (5) deemed to have sensitivity to MUSE -- 2 patients
Groups:
- Daily Sildenafil Citrate: P atients receive oral sildenafil citrate once daily for up to 9 months in the absence of disease progression or unacceptable toxicity. Patients also receive 3 doses of oral sildenafil citrate at least 48 hours apart monthly for up to 18 months. Patients on all three arms will have undergone robotic-assisted laparoscopic surgery. All patients will take part in the questionnaire administration and quality-of-life assessments.
  sildenafil citrate: Given orally
  robotic-assisted laparoscopic surgery: Undergo prostatectomy
  quality-of-life assessment: Ancillary studies
  questionnaire administration: Ancillary studies
Period: Overall Study
Arm/Group | Sildenafil Citrate/Mo+Aprostadil/Day | Sildenafil Citrate Monthly | Daily Sildenafil Citrate
Started | 34 | 35 | 31
Completed | 17 | 19 | 20
Not Completed | 17 | 16 | 11

BASELINE CHARACTERISTICS:
Groups:
- Sildenafil Citrate Monthly Daily Sildenafil Citrate: Patients receive oral sildenafil citrate once daily for up to 9 months in the absence of disease progression or unacceptable toxicity. Patients also receive 3 doses of oral sildenafil citrate at least 48 hours apart monthly for up to 18 months. Patients on all three arms will have undergone robotic-assisted laparoscopic surgery. All patients will take part in the questionnaire administration and quality-of-life assessments.
  sildenafil citrate: Given orally
  robotic-assisted laparoscopic surgery: Undergo prostatectomy
  quality-of-life assessment: Ancillary studies
  questionnaire administration: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Sildenafil Citrate/Mo+Aprostadil/Day | Sildenafil Citrate Monthly | Sildenafil Citrate Monthly Daily Sildenafil Citrate | Total
Number analyzed (Participants) | 34 | 35 | 31 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [53 to 60] | 58 [52 to 61] | 59 [52 to 61] | 58 [53 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 34 | 35 | 31 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 7
  White | 31 | 32 | 25 | 88
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 35 | 31 | 100

OUTCOME MEASURES:

1. Primary Outcome: Potency Rates (Ability to Obtain an Erection Sufficient for Penetration) Without Assistance Compared Between Patients in All Three Arms of the Study at 12 Months
Description: Potency rates (ability to obtain an erection sufficient for penetration) without assistance in those patients receiving maintenance Viagra compared to non-pharmacology controls was compared at 12 months from start of treatment using the fisher's exact test
Time Frame: 12 months following BNS-RAP
Population: These are the patients who remained on treatment for the duration of the 12 months and were evaluable at that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil Citrate/Mo+Aprostadil/Day | Sildenafil Citrate Monthly | Daily Sildenafil Citrate
Number analyzed (Participants) | 17 | 19 | 20
Participants | 13 | 16 | 16
Statistical Analysis 1: Comparison: Sildenafil Citrate/Mo+Aprostadil/Day vs Sildenafil Citrate Monthly vs Daily Sildenafil Citrate; Test type: Equivalence — The equivalence margin that would be possible to detect (had the protocol reached intended accrual) was 20%,; p > 0.1, Fisher Exact — no adjustments were made

2. Secondary Outcome: Potency Rates With or Without Assistance in the Control Group Versus Maintenance MUSE or Maintenance Viagra
Description: Potency rates with or without assistance in the control group versus maintenance MUSE or maintenance Viagra were compared at each of 6 and 18 months
Time Frame: At 6 and 18 months
Population: patients who were evaluated at 6 months, 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil Citrate/Mo+Aprostadil/Day | Sildenafil Citrate Monthly | Daily Sildenafil Citrate
Number analyzed (Participants) | 17 | 19 | 20
Participants
  6 month potency | 10 | 11 | 17
  18 month potency | 14 | 16 | 15
Statistical Analysis 1: Comparison: Sildenafil Citrate/Mo+Aprostadil/Day vs Sildenafil Citrate Monthly vs Daily Sildenafil Citrate; compare percentage of patients potent at 6 and 18 months across pairs of treatment arms (arm I vs arm II, arm I vs arm III, arm II vs arm III); Test type: Other; p > 0.1, Chi-squared — no adjustments done; no adjustments

3. Secondary Outcome: SHIMS-5 Scores in the Control Groups Versus Maintenance MUSE or Maintenance Viagra Groups
Description: Median and range of SHIM scores evaluated at 1, 3, 6, 9, 12, and 18 months. SHIMS-5 is the Sexual Health Inventory for Men, which includes 5 questions that are scored from 1 to 5 each. The total score is obtained by adding all five response scores, and can range from 5 to 25 when all 5 questions are answered. Questions that are left unanswered are scored as a 0, and can result in an overall score lower than 5 (as low as 0). Higher scores are more desirable. A Score of 22-25 = no ED, 17-21=Mild ED, 12-16=Mild to moderate ED, 8-11=Moderate ED, and 5-7 =Severe ED (ED=Erectile Dysfunction). There are no sub-scale scores within this questionnaire.
Time Frame: At 1, 3, 6, 9, 12, and 18 months
Population: patients with shim scores at 1 month
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Sildenafil Citrate/Mo+Aprostadil/Day | Sildenafil Citrate Monthly | Daily Sildenafil Citrate
Number analyzed (Participants) | 16 | 18 | 19
units on a scale
  SHIM score 1 month | 9.5 [1 to 24] | 3 [0 to 25] | 12 [1 to 25]
  SHIM score 3 months: number analyzed (Participants) | 15 | 18 | 19
  SHIM score 3 months | 14 [1 to 21] | 14 [1 to 25] | 18 [1 to 25]
  SHIM score 6 months: number analyzed (Participants) | 15 | 16 | 18
  SHIM score 6 months | 18 [4 to 25] | 18.5 [4 to 25] | 20 [2 to 25]
  SHIM score 9 months: number analyzed (Participants) | 16 | 18 | 18
  SHIM score 9 months | 18.5 [1 to 25] | 17.5 [1 to 25] | 19 [2 to 25]
  SHIM score 12 months: number analyzed (Participants) | 15 | 18 | 19
  SHIM score 12 months | 20 [1 to 25] | 19 [1 to 25] | 18 [3 to 25]
  SHIM score 18 months: number analyzed (Participants) | 16 | 17 | 19
  SHIM score 18 months | 19.5 [1 to 25] | 20 [2 to 25] | 20.5 [2 to 25]
Statistical Analysis 1: Comparison: Sildenafil Citrate/Mo+Aprostadil/Day vs Sildenafil Citrate Monthly vs Daily Sildenafil Citrate; Test type: Other; p > 0.2, ANOVA — no adjustments done

4. Secondary Outcome: Penile Length
Description: measurement of penile length in centimeters
Time Frame: At pre-treatment and 18 months
Population: patients who were willing to have penile measurements taken at baseline
Measure: Median (Full Range); unit: centimeters
Arm/Group | Sildenafil Citrate/Mo+Aprostadil/Day | Sildenafil Citrate Monthly | Daily Sildenafil Citrate
Number analyzed (Participants) | 27 | 26 | 25
centimeters
  Baseline Penile Measurement | 11 [5 to 15] | 12 [6 to 16] | 10.2 [6.4 to 15]
  Month 18 Penile Measurement: number analyzed (Participants) | 19 | 17 | 17
  Month 18 Penile Measurement | 12.5 [8.3 to 14.5] | 11 [3 to 14] | 12 [5.5 to 15.5]
Statistical Analysis 1: Comparison: Sildenafil Citrate/Mo+Aprostadil/Day vs Sildenafil Citrate Monthly vs Daily Sildenafil Citrate; ANOVA test to compare difference of penile length (from baseline to month 18) across arms. calculations are underpowered, as study did not accrue or retain patients as intended, and many patients declined to have measurements taken; Test type: Other; p = 0.08, ANOVA — no adjustments; no adjustments for df; Mean Difference (Final Values) = 0.08

ADVERSE EVENTS:
Time Frame: The time frame was over 1 year.
Description: The drugs that were tested on patients on the three arms are all FDA-approved drugs and were prescribed/provided in doses that were FDA-approved.
Arm/Group | Sildenafil Citrate/Mo+Aprostadil/Day | Sildenafil Citrate Monthly | Daily Sildenafil Citrate
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/31
Other Adverse Events (participants affected / at risk) | 24/34 | 19/35 | 24/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil Citrate/Mo+Aprostadil/Day (N=34) | Sildenafil Citrate Monthly (N=35) | Daily Sildenafil Citrate (N=31)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 7 (7) | 3 (3)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 2 (2) | 2 (6) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 2 (5) | 4 (7)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 1 (1) | 3 (10)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (2) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema trunk (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (2) | 4 (5)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (7) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bladder anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (7) | 9 (29) | 10 (24)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Libido decreased (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Hematuria (Renal and urinary disorders) | 4 (5) | 2 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 1 (1) | 2 (6)
Urinary incontinence (Renal and urinary disorders) | 3 (3) | 3 (8) | 3 (8)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 10 (17) | 2 (2) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 8 (13) | 3 (3) | 2 (2)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (3)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 3 (4) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 8 (27) | 5 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Flushing (Vascular disorders) | 2 (4) | 8 (17) | 5 (12)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
In addition to the fact that the trial was closed mid-way through accrual, nearly half of those that accrued dropped out prior to completing treatment. There is not enough power to make any conclusions regarding any of the aims set forth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes